CLINICAL TRIAL: NCT05249725
Title: Therapeutic Effect of Isogladine Maleate on Small Intestinal Mucosal Injury Associated With NSAIDS in Population
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GSL-LEES-2021-12
Record Dates: First submitted 2022-01-19; First posted 2022-02-22 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: NSAIDs-associated Intestinal Mucosal Injury
Keywords: NSAIDs, intestinal mucosal injury
MeSH Terms: interventions — irsogladine; hydrotalcite

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irsogladine Maleate (Experimental)
  Interventions: Drug: Irsogladine Maleate
- Hydrotalcite (Placebo Comparator)
  Interventions: Drug: Hydrotalcite

INTERVENTIONS:
Drug: Irsogladine Maleate — Orally administration of irsogladine maleate 4mg/day, for 8 weeks.
  Arms: Irsogladine Maleate
Drug: Hydrotalcite — Patients were given 1 g hydrotalcite every morning, afternoon and evening for 8 weeks.
  Arms: Hydrotalcite

SUMMARY:
All patients who met the inclusion criteria and agreed to participate in the study underwent baseline capsule endoscopy. Patients with intestinal mucosal injury detected during the initial capsule endoscopy were randomly divided into isoladin maleate group or magnesium aluminum carbonate control group using computer-generated random numbers. Patients in the isoladine maleate group received 4 mg isoladine maleate (Gesellon, Japan) every morning for 4 weeks (or 8 weeks, duration to be determined); Magnesium aluminum carbonate control group received 1 g magnesium aluminum carbonate every morning, afternoon and evening for 4 weeks (or 8 weeks, course to be determined). After treatment, capsule endoscopy was performed again to evaluate the healing of intestinal mucosa.

DETAILED DESCRIPTION:
In this prospective randomized controlled study, 100 patients with NSAIDS-related intestinal mucosal injury will be enrolled in 10 clinical centers across China from July 2021 to December 2022. All patients who met the inclusion criteria and agreed to participate in the study underwent baseline capsule endoscopy. Patients with intestinal mucosal injury detected during the initial capsule endoscopy were randomly divided into isoladin maleate group or magnesium aluminum carbonate control group using computer-generated random numbers. Patients in the isoladine maleate group received 4 mg isoladine maleate (Gesellon, Japan) every morning for 4 weeks (or 8 weeks, duration to be determined); Magnesium aluminum carbonate control group received 1 g magnesium aluminum carbonate every morning, afternoon and evening for 4 weeks (or 8 weeks, course to be determined). After treatment, capsule endoscopy was performed again to evaluate the healing of intestinal mucosa. Laboratory tests including blood routine, stool routine, and occult blood were performed at the beginning and end of the study. Abdominal symptoms and signs were assessed by two experienced clinicians at week 0, 1, 2, and 4 (8) of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Within 4 weeks before the study, NSAIDs were taken at least once a day with symptoms and signs of abdominal discomfort, such as abdominal pain, abdominal distension and dyspepsia;
2. During the 8-week observation period of the study, NSAIDs will continue to be used in the same protocol (whether to stop NSAIDs during the study remains to be determined);
3. Patients taking antisecretory drugs such as proton pump inhibitors or H2 receptor antagonists and gastric mucosal protectors such as rebapide or tiprexone were eligible;
4. Willing to sign informed consent

Exclusion Criteria:

1. Active gastrointestinal bleeding;
2. Taking more than two NSAIDs, anticoagulants, steroid hormones or prostaglandin derivatives;
3. Have a history of gastrointestinal surgery except appendectomy;
4. Suspected small bowel obstruction;
5. gastroduodenal ulcer;
6. Severe cardiopulmonary diseases (NYHA grade IV cardiac function or respiratory failure);
7. Significant renal impairment (serum creatinine ≥2 mg/dL or glomerular filtration rate GFR<40 mL/min);
8. Liver insufficiency (liver function: total bilirubin >ULN, ASpartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALP) ≥ 2.0 × ULN);
9. Confirmed or suspected combined with malignant tumor;
10. pregnant and lactation women or women who do not exclude the possibility of pregnancy;
11. Drug addicts or alcoholics;
12. Participants in other drug trials within 3 months;
13. The researcher considers it unsuitable for participants

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Number of small intestinal mucosal lesions under capsule endoscopy | 8 weeks
  After 8 weeks of treatment, capsule endoscopy was repeated, and the number of small intestinal mucosal lesions under the microscope decreased by ≥1 or the Lewis score decreased by more than before, which was considered effective.

IPD SHARING:
Plan to Share IPD: Undecided